CLINICAL TRIAL: NCT05792475
Title: Evaluation of TaiHao Breast Ultrasound Diagnosis Software (Plan for Partial Modification of Diagnostic Performance)
Brief Title: Evaluation of TaiHao Breast Ultrasound Diagnosis Software RN-CES Descartes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TaiHao Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TaiHao TVGH2020-07-006AC#1
Record Dates: First submitted 2023-02-10; First posted 2023-03-31 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Define Standard of Truth (SOT) by 3 experts (Other): Three experts A, B, and C independently define standard of truth (SOT) about 108 cases.
  Interventions: Diagnostic Test: Define Standard of Truth (SOT) by Taihao Breast Cancer Diagnostic Software

INTERVENTIONS:
Diagnostic Test: Define Standard of Truth (SOT) by Taihao Breast Cancer Diagnostic Software — TaiHao Breast Cancer Diagnostic Software independently define standard of truth (SOT) about108 cases.

SUMMARY:
A standard of truth "SOT" is determined based on the interpretation results of the case data by interpretation experts, and the SOT is compared with the detection results of this program's function for detecting suspected breast cancer (CADe function). Estimate the detectability of the CADe function by comparing.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20 to 69, including those with and without breast lesions.

Exclusion Criteria:

* Have a pacemaker or prosthetic valve.
* A post-surgery follow-up patient.

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The average performance of the 4 machines, in terms of sensitivity for detecting suspicious breast cancer, is not inferior to Siemens performance. | 1 week
  The average of 4 types of machines (Canon Aplio i800, GE Logiq E10, GE Invenia ABUS, Fuji ARIETTA 60) performance compared to Siemens performance which was submitted to PMDA last time.

SECONDARY OUTCOMES:
The performance of each of the 4 machines, in terms of sensitivity for detecting suspicious breast cancer, is not inferior to Siemens' performance. | 1 week
  Each machine (Canon Aplio i800, GE Logiq E10, GE Invenia ABUS, Fuji ARIETTA 60) performance compared to Siemens performance which was submitted to PMDA last time.

CONTACTS AND LOCATIONS:
Locations (1):
- TaiHao Medical Inc, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT05792475/Prot_000.pdf